CLINICAL TRIAL: NCT04159402
Title: Medical Doctors(Department of Obstetrics and Gynecology)
Brief Title: Dissect Assembly Rules of SPET12 Complex in the Mammalian Sperm
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: A-ER-102-438
Record Dates: First submitted 2019-10-28; First posted 2019-11-12 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2019-11

CONDITIONS: Spermatozoa; Fertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sperm

SUMMARY:
The sperm of the KO mouse shothe investigatorsd severe defects of all found compartments: acrosome, nucleus, midpiece and tail. The investigators also found SEPT12 co-localizes and interact with SEPT1, 2, 4, 6, 7, 10, 11, and 14 in sperm. Interestingly, some of these septins form filaments with SEPT12 in cells. Based on these findings, it is hypothesized that (1) The core complex of SEPT12 filament consists of SEPT12-7-6-2-2-6-7-12; (2) Septin12 mutations, genetic variants, as the investigatorsll as haploinsufficiency disrupt SEPT12 filament and macro-complex; (3) Other SEPT's (e.g. SETP4, SEPT14) are also involved in the functionality of SEPT12; and (4) SEPT12 macro-complex is critical for compartment formation during terminal differentiation of male germ cells. The proposed study is designed to confirm the above hypotheses, to deconstruct mammalian SEPT12 complex, and to elucidate the functional significance of Septin12 mutations. In the proposed study, the investigators will use different methods, including proteomics, immunofluorescence assay, co- immunoprecipitation, pull-down assay, protein domain mapping, and protein complex fractionation to test the above hypothesis. The investigators have created a mouse carrying an important Septin12 mutation. In the proposed study, the investigators plan to knock out Septin14 in the mouse. SEPT14 interacts with SEPT12 and is also predominantly expressed in sperm. The mouse models and research tools could be used to explore the role of septins during spermiogenesis, to deconstruct the SEPT12 complex in the mammalian sperm, and to elucidate the functional significance of the Septin 12 mutations. Our findings may provide novel insight into the pathways human spermatogenesis, and has the potential to lead to development of therapeutic models for male infertility, and design of male contraceptives.

DETAILED DESCRIPTION:
Redundancy and Interchangeability of Septins Septins 3, 4, 5, 6, 11, and 12 have been knocked out in the mouse model. Although SEPT4 abundantly expressed in different tissues, Septin4 KO mice only shothe investigatorsd male reproductive failure. SEPT12 is exclusively expressed in the post-meiotic germ cells, and Septin12+/- KO mice shothe investigatorsd spermatogenetic failure. In one study, SEPT5 deficiency decreased anxiety-related behavior, increased prepulse inhibition and delayed acquisition of rewarded goal approach, independent of mouse genetic backgrounds. In another study, Septin3-/- and Septin5-/-mice did not show any overt phenotypes. Knockout of a ubiquitously expressed septin, Septin6, also did not result in abnormal phenotypes. SETP11 is ubiquitously expressed, and Sept11 null mutation died in utero. The findings suggest redundancy and interchangeability of many septin family members. Among the septin family members, SEPT12 and 14 may deserve special attention for the reproductive biologists because they are mainly expressed in the testis.

ELIGIBILITY:
inclusion criteria:

* All participants signed a written informed consent form.
* Semen samples were obtained by masturbation after 3-5 days of sexual abstinence.

exclusion criteria:

．None

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The participants were clinically diagnosed by semen analysis and further collected the normal human sperm.
Sampling Method: Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2014-08; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Losses of SEPT12, SEPT7, SEPT6, SEPT2 and SEPT4 from the sperm annulus of a SEPT12D197N patient. | 1 day
  Immunofluorescence staining of normal sperm in a fertile control showed signals for SEPT12 . SEPT7, SEPT6, SEPT2 and SEPT4 (red) at the annulus. Also shown are merged fluorescence staining images with the additional staining of the sperm nuclei, as well as merged fluorescence staining images with merged brightfield images (BF merged). Blue color, DAPI stain; BF, brightfield only. Scale bar: 10 µm.

CONTACTS AND LOCATIONS:
Overall Officials: Pao-Lin Kuo, MD, Principal Investigator — Department of Obstetrics and Gynecology, National Cheng Kung University Hospital